CLINICAL TRIAL: NCT06727370
Title: Cognitive Screening in Lung Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 2027
Record Dates: First submitted 2024-11-21; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Lung Disease; NSCLC (Non-small Cell Lung Cancer); SCLC
Keywords: lung cancer; nsclc; sclc; cognitive
MeSH Terms: conditions — Lung Diseases; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients diagnosed with lung cancer: patients diagnosed with lung cancer (both SCLC and NSCLC)

SUMMARY:
This study aims to investigate the occurrence of cancer and adjuvant therapy-related cognitive impairment in patients with both NSCLC and SCLC. The primary endpoint measure will be the presence of cognitive impairment during the first year after enrollment through the administration of a comprehensive neuropsychological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Small-cell and non-small-cell lung cancer (stage I, II, III, IV)
* Age ≥ 18 years
* Patients able to speak and read the local language(s) fluently
* Acceptance and signature of informed consent

Exclusion Criteria:

* Age ≥ 70
* Presence of brain metastases
* Patients with concomitant neurological or psychiatric disorders.
* Patients undergoing brain radiotherapy
* Previous diagnosis of lung cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with lung cancer (both SCLC and NSCLC)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
cognitive impairment | From baseline to 12 months
  It will be the presence of cognitive impairment through the administration of a comprehensive neuropsychological assessment.Patient will complete cognitive evaluation which includes:the Montreal Cognitive Assessment and the Mini-Mental State Examination to assess global cognitive functioning;the Frontal Assessment Battery,the Stroop test color and word test ,and the Verbal Fluency Test for the evaluation of executive function;the Ray Auditory Verbal Learning Test for learning and memory;the forward and backward Digit Span and the Corsi Block-tapping Test for working memory;and the Trail Making Test A & B and the Symbol Digit Modalities Test for attention. Classification will be obtained adopting the criteria proposed by the International Cognition and Cancer Task Force,a test score of 2 SDs or more below the test-specific reference cohort on at least 1 test of a cognitive domain.All test scores were transformed into z-scores to allow the comparison between different measures.

SECONDARY OUTCOMES:
Risk factors on the cognitive profile of lung cancer patients | From baseline to 12 months
  This study will assess the influence of different risk factors on the cognitive profile of lung cancer patients. It will examine the role of psychological symptoms through different self-reported questionnaire: the Functional Assessment of Cancer Therapy - cognition will be administered to assess perceived cognitive impairment, the Beck Depression Inventory II to measure the presence of depressive symptoms, the State-Trait Anxiety Inventory to investigate both state anxiety and trait anxiety, the EORTC-Quality of Life of cancer patient to assess the quality of life and, finally, the Pittsburgh Sleep Quality Index to evaluate sleep quality and disturbances sleep patterns. Finally, the Cognitive Reserve Index questionnaire will be administered to obtain the cognitive reserve level of each patient, and the smoking information obtained through an interview.All the questionnaire scores were transformed into z-scores to allow the comparison between different measures.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy